CLINICAL TRIAL: NCT06142773
Title: Study to Investigate an Association Between Brain Activity and Tidal Volume in Humans (BATMAN) - a Pilot Study
Brief Title: Study to Investigate an Association Between Brain Activity and Tidal Volume in Humans (BATMAN)
Acronym: BATMAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 23-5052
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-01

CONDITIONS: Ventilation Therapy; Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: tidal volume delivered at 6 ml/kg for 3-5 minutes, followed by 12ml/kg for 3-5 minutes (Experimental): The clinical MRI examination will be obtained before commencing with the study protocol. The study protocol will commence once the scheduled MRI scan is finished. The study-related procedures will add 10 minutes after the scheduled MRI scans are finished with two different tidal volumes with maintaining isocapnia and isooxia.
  Study procedure: tidal volume delivered at 6 ml/kg for 5 minutes, followed by 12ml/kg for 5 minutes
  Interventions: Device: Tidal Volume set on ventilator
- Group 2: tidal volume delivered at 12 ml/kg for 3-5 minutes, followed by 6ml/kg for 3-5 minutes (Active Comparator): The clinical MRI examination will be obtained before commencing with the study protocol. The study protocol will commence once the scheduled MRI scan is finished. The study-related procedures will add 10 minutes after the scheduled MRI scans are finished with two different tidal volumes with maintaining isocapnia and isooxia.
  Study procedure: tidal volume delivered at 12 ml/kg for 5 minutes, followed by 6ml/kg for 5 minutes
  Interventions: Device: Tidal Volume set on ventilator

INTERVENTIONS:
Device: Tidal Volume set on ventilator — Mechanically ventilated patients who are undergoing MRI examinations under general anesthesia in isocapnic and isoxic conditions will have brain activity investigated under two different tidal volumes, 6 ml/kg and 12 ml/kg applied for 3-5 minutes.

SUMMARY:
The communication between the lungs and the brain has drawn a lot of attention recently. Animal studies have shown that the breathing cycle is coupled with brain activity, showing that the greater the volume of air delivered to the lungs via a breathing machine greater the brain activity and also the greater the injury to the brain cells.

There is no study in humans that investigates the physiological communication between the volume of air delivered to the lungs and brain activity. This is important because really sick patients receive breathing assistance using breathing machines to keep their oxygen levels within a normal range. Although these machines are life-saving tools, they might result in brain cell injury, leading to cognitive impairment. So, establishing the existence of a physiological communication between the volume of air delivered using these breathing machines and brain activity is the first step to investigating therapies to prevent brain cell injury due to the use of breathing machines to assist breathing.

DETAILED DESCRIPTION:
Demonstration of a physiological relationship between tidal volume set on the ventilator and hippocampal activity measured as changes in blood-oxygenation level-dependent (BOLD) in the regions of interest (ROIs). The results from this pilot study might assist in creating the foundation for explaining the mechanism of action of ventilation-associated brain injury.

Mechanically ventilated patients who are undergoing MRI examinations under general anesthesia in isocapnic and isoxic conditions will have brain activity investigated under two different tidal volumes, 6 ml/kg and 12 ml/kg applied for 3-5 minutes. Positive end-expiratory pressure will be adjusted to maintain plateau pressure <30 cm H2O.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled to undergo an MRI scan of their head under general anesthesia
2. Age > 18 years

Exclusion Criteria:

1. Stroke, and/or brain tumor in the regions of interest that has not been diagnosed before the MRI scan
2. Previous medical history of dementia
3. Previous medical history of brain surgery
4. Acute or chronic spinal cord Injury
5. Previous Vagotomy
6. Phrenic nerve injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
establish a correlation between the tidal volume delivered and changes in the blood-oxygenation level-dependent (BOLD) on regions of interest (ROIs) during an MRI scan. | 10 minutes
  correlation between the tidal volume delivered and changes in the blood-oxygenation level-dependent (BOLD) on regions of interest (ROIs)

SECONDARY OUTCOMES:
establish whether the changes in BOLD signal in multiple ROIs correlate with changes in tidal volume via a multi-correlation analysis (independent component analysis) | 10 minutes
  establish whether the changes in BOLD signal in multiple ROIs correlate with changes in tidal volume via a multi-correlation analysis

CONTACTS AND LOCATIONS:
Overall Officials: Ewan Goligher, MD, Principal Investigator — University Health Networ
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada